CLINICAL TRIAL: NCT00353249
Title: Cognitive Behavioral Therapy for Homeless Women With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Cognitive Behavioral Therapy for Post-Traumatic Stress Disorder in Homeless Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Suzanne Wenzel, RAND Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH076099 (NIH); R34MH076099 (NIH); DSIR 82-SEMS
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Cognitive Behavioral Therapy; CBT; Homeless Women
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

ARMS (2):
- 1 (Experimental): Participants will receive adapted cognitive behavioral therapy treatment
  Interventions: Behavioral: Adapted cognitive behavioral therapy (CBT)
- 2 (No Intervention): Participants will receive no treatment for the course of the study; they will be offered courtesy PTSD 5 weeks after the experimental intervention.

INTERVENTIONS:
Behavioral: Adapted cognitive behavioral therapy (CBT) — Adapted CBT is a group treatment for PTSD and will occur two times per week for 4 weeks. The sessions will last 90-minutes and will be led by a therapist and co-therapist.
  Arms: 1

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy in treating post-traumatic stress disorder in homeless women.

DETAILED DESCRIPTION:
Exposure to traumatic events may lead to mental health problems, such as post-traumatic stress disorder (PTSD). PTSD is a type of anxiety disorder that is characterized by the presence of persistent frightening thoughts and memories of the traumatic event. Additionally, people with PTSD often feel emotionally numb, and they may experience sleep problems or be easily startled. Homeless people, in particular, are at risk for experiencing a variety of traumas. Homeless women tend to experience more traumatic events and develop PTSD at higher rates than housed women. Although effective treatments for PTSD are available, homeless women are unlikely to seek them out. There is a need for PTSD treatment approaches that are specifically designed for these women. This study will develop a cognitive-behavioral therapy treatment that will be adapted to best serve the needs of homeless women. The study will then determine the therapy's effectiveness in treating a group of homeless women with PTSD.

This study will consist of three phases. The first phase will be used to gather and analyze information about PTSD in homeless women and methods of treating the disorder in this population. Focus groups consisting of homeless women, shelter directors, case managers, and mental health service providers will be used to obtain the necessary information. Phase two of this study will consist of developing an adaptation of an existing PTSD treatment manual to make it relevant to the lives of homeless women. The third and final phase of this study will recruit 32 homeless women with symptoms of PTSD, and who did not participate in either of the first two phases of the study. Participants in this 4-week study will be randomly assigned to receive either the adapted cognitive behavioral therapy treatment or no treatment at all (assessment-only). The treatment group will attend twice weekly sessions for a total of 4 weeks. All participants will be evaluated immediately prior to the start of treatment and 1 week after treatment ends. Outcomes will include PTSD symptoms and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Sub-diagnostic threshold PTSD symptoms
* Currently resides in a transitional homeless shelter in Los Angeles County
* Trauma that is related to PTSD symptoms occurred at least 1 month prior to study entry
* Understands, speaks, and reads English
* Planned departure date from the shelter is at least 1 month after study entry

Exclusion Criteria:

* Significant cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | Measured at Week 4
Depression symptoms | Measured at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Wenzel, PhD, Principal Investigator — RAND
Locations (1):
- Los Angeles County, California, United States